CLINICAL TRIAL: NCT04756297
Title: Lung Ultrasound for Prediction of Bronchopulmonary Dysplasia in Extremely Preterm Neonates: A Prospective Diagnostic Cohort Study
Brief Title: Lung Ultrasound for Prediction of Bronchopulmonary Dysplasia
Status: Completed | Type: Observational
Sponsor: Adel Mohamed (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); Health Sciences Centre, Winnipeg, Manitoba (Other)
Responsible Party: Sponsor-Investigator, Adel Mohamed, Assistant professor of Paediarics, Mount Sinai Hospital, Canada
Organization: Mount Sinai Hospital, Canada (Other)
Other Study IDs: 19-0072-E
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Bronchopulmonary Dysplasia (BPD)
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extreme preterm infants (GA ≤ 28+6 weeks) are at high risk for bronchopulmonary dysplasia (BPD) that has been associated with significant long-term impairment. Lung ultrasound score (LUSs) has the potential to early identify infants at high risk of developing BPD who may benefit from early intervention.

Aim: To assess if LUS score can be utilized to predict the development of BPD in infants born at ≤ 28+6 weeks, early in their postnatal course, when the disease is likely to be most amenable to therapeutic intervention.

DETAILED DESCRIPTION:
Background and Importance: Despite advances in neonatal care and improved survival among immature infants, bronchopulmonary dysplasia (BPD) remained a serious complication among preterm neonates born at <29 weeks' gestational age. A variety of therapies including antenatal steroid, surfactant administration, high-frequency ventilation, postnatal steroid (systemic and inhaled), and vitamin A supplementation have been studied as means to prevent BPD. Ideally, interventional studies aim to prevent or reduce BPD should include criteria for selecting infants at highest risk for BPD while excluding infants at low risk. Recently, Lung ultrasound severity score (LUSs) has shown in few studies to be a promising tool for assessing lung aeration and for early prediction of preterm infants with evolving BPD. These studies have a major limitation as it includes infants at low risk for BPD (> 28 weeks gestational age). In this study, we will assess the accuracy of LUSs for early identification BPD among extreme preterm infants born at <29 weeks' GA.

Study procedure In this prospective observational study, our aim is to recruit a large cohort of extreme premature neonates (born at ≤ 28+6 weeks gestational age), and sequentially perform an "early-diagnostic assessments "on day 3 of age. Subsequent LUS assessment will be performed at 7 days (+/- 1 day) of age and the third LUS assessment will be at 14 (+/-2 days of age). Assessment will be done in the same manner as described by Cattarossi et.al. Basically, each lung will be divided into 3 zones (upper anterior, lower anterior, and lateral) and will be examined using a L20 linear probe to perform a longitudinal lung scan (Fig 1). Additionally, we will score each zone (score 0-to 3 points) according to the modified LUS score by Brat et.al [20]. Based on the LUS pattern in each lung zone the total score can range from 0 to 18 for the 6 zones of both lungs. As summarized in figure 2 the LUS score will include signs that can be used to diagnose TTN, RDS or identify early changes of BPD.

We will record this data for babies enrolled in the study, along with their relevant medical data. At the end of this study, we will divide the cohort into those who developed BPD and those who did not as per currently used standard criteria and will compare the results of new LUS severity score obtained at earlier time points. Prediction models will be created including variables associated with BPD development at each time point with and without inclusion of lung US severity score.

Regarding LUS assessment a Zonare Ultrasound machine (Z.One PRO ultrasound) with a high-frequency (L20-5) linear probe will be used. This high-frequency probe gives excellent resolution and adequate penetration in these small infants. We decided to start LUS scanning at day 3 of age as most of these babies are at risk for intraventricular hemorrhage and minimal handling especially during the first 3 days is highly recommended.

All LUS assessments will be undertaken at the same time using a standard aseptic technique and without too much handling of the infants. Approval will be obtained from the Research Ethics Board (REB) at Sinai Health System and Health sciences Centre-Winnipeg. Parents will be approached for consent before enrollment.

ELIGIBILITY:
Inclusion Criteria:

GA ≤ 28+6 weeks Admitted to the NICU at Mount Sinai Hospital or Health sciences Centre-Winnipeg consent obtained.

Exclusion Criteria:

Infants who are born at > 28 weeks GA, or have congenital or chromosomal abnormalities, or parents declined consent will be excluded.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants who are born at GA ≤ 28+6 weeks will be enrolled in the study after obtaining REB approval and parents' consent.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Assess accuracy of LUSs for early identification of BPD in extreme preterm infants | 2 weeks after birth
  The primary outcome of this study is to assess predictive characteristics of LUS score: Sensitivity, specificity, positive and negative predictive value, likelihood ratio and c-statistics of LUS score. Assessment of BPD at 36 weeks will be done as per currently used standard criteria for BPD.
  The primary outcome of this study is to assess predictive characteristics of LUS score: Sensitivity, specificity, positive and negative predictive value, likelihood ratio and c-statistics of LUS score. Assessment of BPD at 36 weeks will be done as per currently used standard criteria for BPD.
  LUS will be conducted at D3, 7 and 14 of life

SECONDARY OUTCOMES:
Assess predictive characteristics of LUS score integration in clinical variables derived model to see which model has higher predictive characteristics | 2 WEEKS
  Different predictive models will be constructed to identify which model best predict BPD

CONTACTS AND LOCATIONS:
Overall Officials: Prakesh Shah, MD, Study Chair — Mount Sinai Hospital- Toronto, ON, Canada
Locations (2):
- Canada (2):
  - Health Sciences Centre, Winnipeg, Manitoba
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Mohamed A, Mohsen N, Diambomba Y, Lashin A, Louis D, Elsayed Y, Shah PS. Lung Ultrasound for Prediction of Bronchopulmonary Dysplasia in Extreme Preterm Neonates: A Prospective Diagnostic Cohort Study. J Pediatr. 2021 Nov;238:187-192.e2. doi: 10.1016/j.jpeds.2021.06.079. Epub 2021 Jul 6. PMID 34237347